CLINICAL TRIAL: NCT04526171
Title: Vaparshun Improving Toilet Use in Rural India (The 5 Star Toilet Campaign)
Brief Title: Vaparshun Improving Toilet Use in Rural India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation of India (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Deepak Saxena, Professor, Public Health Foundation of India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHFindia
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Behavior
Keywords: sanitation; toilet; behavior; evaluation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The study was a cluster-randomised trial with 47 intervention and 47 control clusters, with a baseline and an endline survey conducted in the district of Bhavnagar, Gujarat, India. Briefly, 94 villages were randomised to intervention or control groups. We carried out a household census and from this we selected 10 households with a functional 'government' toilet for a baseline and 30 for follow up at endline using random sampling from the census list for each village. Outcomes were measured as the proportion of households where all members were reported to use the toilet and the overall usage of toilets by individuals, employing a standard questionnaire.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaparshun (Experimental): In intervention clusters, two full day events, with a gap of 4 weeks between the two events, were organized at cluster level. Eligible households with a government or contract tor built toilet were invited to enroll for a toilet makeover. Intervention activities, delivered at cluster level, included films on toilet improvement, comfort and convenience of toile use, addressing pit filling anxiety and celebrating proud toilet owners by providing certificates and acknowledging them during the events.
  Interventions: Behavioral: Vaparshun
- Control Arm (No Intervention): No intervention was delivered to clusters in the control arm.

INTERVENTIONS:
Behavioral: Vaparshun — Participants in the intervention clusters were encouraged to improve their existing toilets.
  Other Names: 5 Star Toilet Campaign
  Arms: Vaparshun

SUMMARY:
Vaparshun intervention aimed to inspire the target audience to use a toilet. It aimed to revalue their toilets by recognizing that they provide benefits associated with the motives of hoard, create, convenience (comfort) and affiliation, and provide a reward pathway for transitioning to a new toilet use routine.

DETAILED DESCRIPTION:
Our intervention consists of four different streams of activity. The outcome is that family members and men improve and use their contractor-built toilets. The activities are listed below.

1. Create Motive:

   Toilet Makeover: Conduct a lottery and perform makeovers of select government built toilets in the village, with the involvement of the community. Demonstrate improvements in comfort (light, space, ventilation, latrine chair/handle) and aesthetics (stencil painting of door and walls).

   Challenge/Opportunity: Many of the 'contractor' toilets are built with low engagement from family members and are uncomfortable to use. People are left with toilets they are not proud of or engaged with.

   Insight (from 'makeover' trial): If families invest in creating an attractive toilet they are be more likely adopt and use them.

   Inputs: Materials for the physical and aesthetic improvement of a toilet, manuals for conducting the community event.

   Outputs: Greater engagement with, and pride in, the toilet after makeover; others in the village inspired to conduct their own makeover. Those who use the upgraded toilet find it a more comfortable experience than they had expected causing reinforcement learning.
2. Hoard motive:

   Pit Emptying Demo and Pit Filling Estimation Demo" A community event-based discussion of the 'real' aspects related to pit filling/emptying designed to graphically overcome their perceptual barriers (e.g., squeezing a watermelon to show how little material there is in faeces).

   Challenge/Opportunity: People over-estimate the speed at which a pit fills and are uncertain about the emptying process. Therefore they hoard the 'limited' pit space by using the toilet only partially.

   Insight from FR: There are gaps between perception and reality which can be addressed. For example; water doesn't stay in the pit but seeps into the soil, faeces are composed mainly of water, decomposition reduces volume, compost doesn't smell and twin pits can be used interchangeably forever.

   Inputs: Films and 'emo-demos' (emotional demonstrations). Outputs: Participants are less anxious about pit filling and emptying.
3. Affiliation/convenience motives:

   Community Motivational Events: Small and large community events such as street plays, films, posters and pledging activities to bring alive convenience/comfort motives by amplifying problems associated with OD and rewards of using toilets; use of affiliation through testimonials films, posters, village maps, etc.

   Challenge/Opportunity: Even if the barriers around pits and toilet comfort are addressed, it may still not be enough to motivate men with entrenched habits of OD to start using toilets.

   Insights: Convenience/comfort can be a powerful drive for toilet usage. Those who use toilets in the village (women, children and elderly) find it is much more convenient and therefore do not return to OD. However, men who are non-users may not have experienced this and need to be convinced. Affiliation can be another strong drive for toilet usage. It is possible to exploit the emerging norms of toilet use and encourage men 'not to be left behind'.

   Inputs: Scripts, props, invitations, loud hailers, audio-visual equipment, etc. Outputs: Men use toilets because they 'get' how convenient they are, and so as not to be 'left behind'.
4. Transition to a new toilet use This would include testimonial videos of toilet users and toilet board of household members who improved their toilets. Providing certificate to households who improved their toilets.

Challenge/Opportunity: Those who use toilets for a specific period tend to stick with the habit; however, some people, especially men, do not try out the toilet or find the first experience unpleasant.

Insight: Reward the use of toilets for a specific period so new habits can form.

Inputs: Stimuli and nudges. Outputs: The entire family, especially men, form the habit of using a toilet.

In addition, village authorities will also be recruited to support delivery of the intervention.

ELIGIBILITY:
Inclusion Criteria:

- Households with a functional government or contractor built toilet.

Exclusion Criteria:

* Households with self built toilet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2483 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of households where all members above the age of 5 years were reported to use the toilet the last time they defecated. | A gap of 6 weeks was maintained between campaign roll out and endline data collection
  The survey was addressed to one adult respondent per household, preferably the male or female household head

SECONDARY OUTCOMES:
Exposure to the intervention | Six weeks post intervention delivery
  Proportion of population in intervention arm that reports attending intervention events
Perceptions related to toilet use | Six weeks post intervention delivery
  Agreement with statements reflecting important campaign messages such as "Toilets are not just for women; men should use them too", "A smart person is one who uses a toilet", or (phrased negatively) "Toilet pits fill quickly if too many people in the household use them"

CONTACTS AND LOCATIONS:
Overall Officials: Deepak o Saxena, PhD, Principal Investigator — IIPHG
Locations (1):
- Indian Institute of Public Health/ Public Health Foundation of India, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol, SAP
Time Frame: Now.
Access Criteria: Unlimited.
URL: http://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/Q3P4WX

REFERENCES:
- [Derived] Schmidt WP, Chauhan K, Bhavsar P, Yasobant S, Patwardhan V, Aunger R, Mavalankar D, Saxena D, Curtis V. Cluster-randomised trial to test the effect of a behaviour change intervention on toilet use in rural India: results and methodological considerations. BMC Public Health. 2020 Sep 11;20(1):1389. doi: 10.1186/s12889-020-09501-y. PMID 32917160
- See also: Report of the impact evaluation — http://www.3ieimpact.org/sites/default/files/2020-02/IE105-TW14.1002-5-star-toilet-Gujarat.pdf
- Available data/document: Individual Participant Data Set — https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/Q3P4WX

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04526171/Prot_SAP_000.pdf